CLINICAL TRIAL: NCT03873324
Title: One Centre Single Ascending Dose and Double Blind Multiple Ascending Dose, Safety and Pharmacokinetics Phase I Study of CPL500036 Compound in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of CPL500036 Compound in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 01PDE2018
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only PART B will be double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPL500036 (Experimental): PART A: 7 cohorts are to receive single dose of IMP. Each participant is to take single dose of IMP. There is to be dose escalation between cohorts.
  PART B: 4 cohorts are to receive multiple dose of IMP. Each participant is to take IMP once daily for 14 days. There is to be dose escalation between cohorts.
  Interventions: Drug: CPL500036 compound
- Placebo (Placebo Comparator): PART B: 2 Participants from 4 cohorts (total of 8 people) are to receive masking placebo capsules once daily for 14 days. There is to be dose escalation between cohorts. Participants are to be randomized within cohorts.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPL500036 compound — IMP is a capsule with CPL500036 as an Active Pharmaceutical Ingredient (API).
  Arms: CPL500036
Drug: Placebo — matching placebo capsules
  Arms: Placebo

SUMMARY:
The planned study is to determine the safety and pharmacokinetic properties of CPL500036 compound after single and multiple (two weeks) administration in healthy volunteers.

DETAILED DESCRIPTION:
This is to be one-centre, single ascending dose and double-blind multiple ascending dose two part study of CPL500036 compound in healthy volunteers.

PART A is a single dose, open-label part with CPL500036 compound administered with dose escalation between cohorts.

PART B is a multiple, double-blind part with CPL500036 compound administered for 14 days with dose escalation between cohorts. Participants in this part are to be randomized to receive Investigational Medicinal Product (IMP) or placebo in 3:1 ratio.

Safety and pharmacokinetic properties of CPL500036 compound is to be determined following different doses in single oral IMP administration in PART A and different doses of IMP administered orally for two weeks in PART B.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian female or male,
* Age: 18-55 years old, inclusive,
* Body-mass index (BMI): ≥18.5 kg/m^2 and <29.9 kg/m^2,
* Non-smoker and nonuser of tobacco products for at least 3 months before screening,
* Physical examination without any clinically relevant abnormality,
* Laboratory values not clinically significant,
* Volunteer (or his/her partner) of childbearing potential willingness to use acceptable forms of contraception.

Exclusion Criteria:

* Known allergy or hypersensitivity to other drugs similar in structure or class to CPL500036 compound, or to any excipients of the formulation,
* Any known significant current or past acute or chronic disease or condition,
* Participation in other clinical trial within 90 days preceding the screening,
* Blood drawn within 30 days prior to inclusion to the study (more or equal to 300mL),
* Positive results from pregnancy test for female participants,
* Lactation in women participants,
* Hypotension or hypertension in medical history,
* Long QT interval syndrome or is under the treatment with antiarrhythmic drugs,
* Narcotic, alcohol addiction or abuse,
* Participant who adhere to a special diet (e.g. low calories, vegetarian).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) or administration of the maximum dose provided in the protocol after single and multiple oral administration of IMP. | up to 24 hours after single administration of IMP in PART A and up to 24 hours after the last IMP administration in PART B
  MTD is defined as the highest dose for which no more than 1 of the 6 treated volunteers (less than 1/3) exhibits dose limiting toxicity (DLT).
Safety and tolerability of IMP after single and multiple oral administration based on laboratory values, vital signs, ECG, physical examinations and Adverse Events monitoring. | up to 14 days in PART A and up to 28 days in PART B of the study
  Participants are to be closely observed to assure maximal safety and to collect occurrence of all adverse events. All participants are to be monitored for clinically relevant changes in physical examination, vital signs, 12-lead ECG assessment and deviations from normal in clinical laboratory results (complete blood count, blood chemistry, urinalysis). To follow-up on all study participants telephone calls with a request for information regarding their health condition are to be made.

SECONDARY OUTCOMES:
Cmax - maximum CPL500036 plasma concentration | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  The maximum concentration of the CPL500036 compound in plasma after IMP administration, obtained directly from the measured concentrations.
AUC(0-72) - area under the plasma concentration - time curve from time 0 to 72h after IMP administration for CPL500036 | up to 72 hours after administration of IMP in PART A
  The AUC(0-72) is a measure of total plasma exposure to the drug from time point zero to 72 hours after IMP administration.
AUC(0-24) - area under the plasma concentration - time curve from time 0 to 24h after IMP administration for CPL500036 | up to 24 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 and 14 in PART B
  The AUC(0-24) is a measure of total plasma exposure to the drug from time point zero to 24 hours after IMP administration.
AUC(0-inf) - area under the plasma concentration - time curve from time 0 to infinity time for CPL500036 | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  The AUC(0-inf) is a measure of total plasma exposure to the drug from time point zero extrapolated to infinity.
Tmax - time to reach maximum CPL500036 concentration | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  The Tmax is time to reach the maximum plasma concentration (Cmax), obtained directly from the actual sampling times.
Kel - terminal elimination rate constant | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  Kel is to be estimated via linear regression of time versus log of concentration.
T1/2 - The plasma elimination half-life for CPL500036 compound | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  T1/2 is to be calculated as 0.693/Kel.
C (1,t) - CPL500036 concentration | Determined on Day 2, 3, 4, 5, 6, 8, 9, 10, 11, 12 and 13 in PART B.
  The concentration of CPL500036 on day t before product administration.
C (Tmax, t) - CPL500036 concentration | Determined on Day 2, 3, 4, 5, 6, 8, 9, 10, 11, 12 and 13 in PART B.
  The concentration on day t measured on time Tmax which was calculated in PART A of the study.
Amount of CPL500036 in each urine collection sample | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  It is to be calculated as CPL500036 concentration in urine sample times volume of urine collection.
Ae - total amount of CPL500036 excreted in urine | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  Ae is to be calculated as asymptote of the plot of the cumulative amount of drug excreted after each collection interval plotted against the median of the collection interval.
Clr - renal clearance | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  Clr is to be calculated by linear least squares regression analysis on semi-logarithmic transformed data (CLr = excretion rate/C).
Excretion rate | up to 72 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 7 in PART B and up to 72 hours after the last IMP administration on Day 14 in PART B
  Excretion rate calculated as = CLr/V x Dose x exp(-kt)

CONTACTS AND LOCATIONS:
Locations (1):
- BioResearch Group Sp. z o.o., Kajetany, Nadarzyn, Poland